CLINICAL TRIAL: NCT06959693
Title: mFOLFOX and Cetuximab - β With or Without Envafolimab for MSS, RAS/BRAF Wild - Type Advanced Unresectable CRC: Prospective, Randomized, Controlled Phase Ⅱ/Ⅲ Trial
Brief Title: A Clinical Study to Evaluate the Efficacy and Safety of Envafolimab Combined With Cetuxima-βand mFOLFOX6 in Patients With MSS, RAS/BRAF Wild-Type Metastatic Colorectal Cancer (mCRC)
Status: Not yet recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Rui-hua Xu, MD, PhD, President and Professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SMA CRC 005
Record Dates: First submitted 2025-04-28; First posted 2025-05-06 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-04

CONDITIONS: Metastatic Colorectal Cancer (CRC)
MeSH Terms: conditions — Colorectal Neoplasms | interventions — envafolimab

STUDY DESIGN:
Intervention Model Description: Experimental Arm: Cetuximab β + mFOLFOX6 + Envafolimab • Induction Phase (12 cycles): o Patients receive cetuximab β + mFOLFOX6 + envafolimab. o Patients who achieve CR/PR/SD (no disease progression) after 12 cycles proceed to the maintenance phase. • Maintenance Phase: o Cetuximab β + 5-FU + envafolimab Control Arm: Cetuximab β + mFOLFOX6 • Induction Phase (12 cycles): o Patients receive cetuximab β + mFOLFOX6. o Patients who achieve CR/PR/SD (no disease progression) after 12 cycles proceed to the maintenance phase. • Maintenance Phase: o Cetuximab β + 5-FU
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Envafolimab combining with Cetuximab -β and mFOLFOX6 (Experimental)
  Interventions: Drug: Cetuxima-β; Drug: Envafolimab; Drug: mFOLFOX6
- Cetuximab -β and mFOLFOX6 (Active Comparator)
  Interventions: Drug: Cetuxima-β; Drug: mFOLFOX6

INTERVENTIONS:
Drug: Cetuxima-β — 500 mg/m², initial intravenous infusion (IV)>120 min, subsequent IV >60 min , D1，every 2 weeks
Drug: Envafolimab — a single fixed dose of 200 mg, subcutaneous injection(SC), every 2 weeks (Day 1 of each cycle [D1])
  Arms: Envafolimab combining with Cetuximab -β and mFOLFOX6
Drug: mFOLFOX6 — Oxaliplatin 85 mg/m² , IV, over 120 min, Day 1; Leucovorin 400 mg/m² (or Calcium Folinate 200 mg/m²), IV, over 120 min, D1; 5-FU 400 mg/m² , bolus injection, followed by 1200 mg/(m²·d) continuous IV for 2 days (total dose 2400 mg/m² over 46 - 48 hours)

SUMMARY:
This is a prospective randomized controlled Phase Ⅱ/Ⅲ Clinical study to evaluate the clinical efficacy and safety of Envafolimab combining with Cetuximab -β and mFOLFOX6 in Patients With MSS, RAS/BRAF Wild-Type Metastatic Colorectal Cancer (mCRC)

DETAILED DESCRIPTION:
Patients diagnosed with unresectable, microsatellite - stable (MSS), RAS/BRAF wild - type metastatic colorectal adenocarcinoma who have not received prior systemic anti-neoplastic therapy for metastatic or recurrent lesions will be included in this study.

In the Phase II study, approximately 186 patients will be enrolled, with 93 assigned to the experimental group and 93 to the control group. In the Phase III study, around 404 patients will be recruited, with 202 allocated to the experimental group and 202 to the control group.

Eligible patients will undergo a screening period of up to 28 days, followed by a treatment period consisting of 2 - week cycles for a maximum duration of 2 years. Subsequently, a follow - up period will be implemented, which includes a safety follow - up and survival follow - ups conducted every 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients are eligible for the study if they meet all of the following criteria:

  1. Prior to enrollment, the participant is required to sign a written informed consent form.
  2. Participants should be above 18 years，regardless of gender.
  3. Histopathologically confirmed untreated advanced colorectal adenocarcinoma.
  4. Tumors with RAS (KRAS, NRAS, HRAS) and BRAF wild-type, MSS phenotype, excluding appendiceal or anal cancer. All listed codons must be wild-type: KRAS: Exons 2, 3, 4 (Codons 12, 13, 59, 61, 117, 146) ; NRAS: Exons 2, 3, 4 (Codons 12, 13, 59, 61, 117, 146)
  5. Imaging (enhanced CT/MRI/PET-CT) confirms advanced/metastatic colorectal cancer with measurable lesions according to RECIST v1.1.
  6. No prior systemic therapy for advanced/metastatic colorectal cancer, including chemotherapy, EGFR inhibitors (cetuximab, panitumumab), VEGF inhibitors (bevacizumab), and immune checkpoint inhibitors (anti-PD-1/PD-L1/CTLA-4). Adjuvant/neoadjuvant chemotherapy within 6 months before recurrence/metastasis is considered first-line therapy.
  7. ECOG PS score 0-1.
  8. Expected survival >12 weeks.
  9. Adequate organ function (without blood component or growth factor use within 14 days):

     Hematology:Neutrophils ≥1.5×10⁹/L, platelets ≥100×10⁹/L, hemoglobin ≥90 g/L. Liver/kidney function: SCr ≤1.5×ULN or creatinine clearance ≥50 ml/min, TBIL ≤1.5×ULN, AST/ALT ≤2.5×ULN (≤5×ULN if due to liver metastasis), urine protein <2+ (≤1g/24h if ≥2+).
  10. Normal coagulation, no active bleeding/thrombosis: INR ≤1.5×ULN, APTT ≤1.5×ULN, PT ≤1.5×ULN.
  11. Non-surgically sterile women of childbearing potential must use contraception during and 3 months after treatment; serum/urine HCG negative within 7 days before enrollment; not breastfeeding. Non-surgically sterile men must use contraception with partners during and 3 months after treatment.
  12. Willing participant with good compliance for safety and survival follow-up.

      Exclusion Criteria:

      -
* Patients will be excluded from the study if they meet any of the following exclusion criteria:

  1. Other malignancies in the past or current (excluding cured basal cell carcinoma or cervical carcinoma in situ).
  2. Current duodenal ulcer, ulcerative colitis, intestinal obstruction, or other GI conditions that may cause bleeding or perforation, as judged by the investigator.
  3. Patients with symptomatic pleural, peritoneal, or pericardial effusions requiring treatment.
  4. History of allergy to monoclonal proteins or any component of the study drugs.
  5. Oral traditional Chinese medicine, immunomodulators within 2 weeks, or radiotherapy within 4 weeks before treatment.
  6. Thyroid dysfunction that is uncontrolled by medication.
  7. Uncontrolled hypertension despite receiving optimal treatment (systolic BP>150 mmHg or diastolic BP>90 mmHg).
  8. Uncontrolled cardiac conditions: (1) NYHA Class II+ heart failure; (2) unstable angina; (3) myocardial infarction within 1 year; (4) clinically significant arrhythmias requiring treatment.
  9. Active autoimmune disease or a history of such diseases.
  10. Immunosuppressants, systemic, or absorbable topical steroids for immunosuppression (>10 mg/day prednisone or equivalent) within 2 weeks before enrollment.
  11. CNS metastases.
  12. Active infection or unexplained fever>38.5°C during screening or before first dose (tumor-related fever is acceptable).
  13. History or current evidence of pulmonary fibrosis, interstitial pneumonia, pneumoconiosis, radiation pneumonitis, drug-induced pneumonia, or severe pulmonary dysfunction.
  14. Congenital or acquired immunodeficiency, such as HIV infection, or active hepatitis (elevated transaminases not meeting inclusion criteria, HBV DNA≥1000 IU/ml, HCV RNA≥1000 IU/ml).
  15. Live vaccine administration within 4 weeks before first dose or planned during the study.
  16. History of psychiatric drug abuse, alcoholism, or drug addiction.
  17. Pregnant or breastfeeding women, or those planning pregnancy during the trial.
  18. Any other factor that may lead to premature study discontinuation, as judged by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 590 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2028-09-30 (Estimated); Study Completion 2030-06-30 (Estimated)

PRIMARY OUTCOMES:
Progressin Free Survival，PFS | Time Frame: from the first dose until firstly confirmed and recorded disease progression or death (whichever occurs earlier),assessed up to 3 years
  Progression-free survival based on RECIST v1.1

SECONDARY OUTCOMES:
OS，Overall survival | from the date of first dose unitl the date of death from any cause，assessed up to 3 years
ORR， Objective response | up to 3 years
  Objective response rate based on RECIST v1.1
DCR， Disease control rate | up to 1 year
  the proportion of patients with the best overall response of CR, PR, or stable disease (SD)
NED Rate， No Evidence of Disease Rate | up to 3 years
  The proportion of participants with no evidence of disease after treatment, as determined by current assessments (pathological, imaging, and molecular biology). NED includes complete response (CR), R0 resection, or other local treatments, such as radiofrequency, microwave, or cryoablation (which can be combined with surgery), that eliminate the tumor.
Safety(Adverse Event (AE) Incidence) | up to 3 years
  Adverse Event (AE) Incidence

CONTACTS AND LOCATIONS:
Locations (1):
- Medical Oncology,Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China